CLINICAL TRIAL: NCT01840735
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Single Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of GS-5737 in Subjects With Cystic Fibrosis
Brief Title: Phase 1b Safety, Tolerability, and PK Study to Assess GS-5737 in Subjects With CF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-234-0117
Record Dates: First submitted 2013-04-15; First posted 2013-04-26 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Cystic Fibrosis
Keywords: CF; Cystic Fibrosis; PK
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GS-5737 (Active Comparator): The GS-5737 85 μg dose is contained in 4 mL of 10 mM citrate buffer, pH 5.0 in 2.8% (w/v) saline.
  Interventions: Drug: GS-5737
- Placebo (Placebo Comparator): The vehicle (placebo) control contains 10 mM citrate buffer, pH 5.0 in 2.8% (w/v) saline in 4 mL.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-5737
  Arms: GS-5737
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will determine the safety, tolerability, and pharmacokinetics of a single dose of GS-5737 administered with a 2.8% saline solution vehicle in adult subjects with CF.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ≥ 18 years of age, at Screening
* Diagnosis of CF as determined by the 1997 CF Consensus Conference criteria, with at least 1 of the following: Documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test OR Abnormal nasal transepithelial potential difference (NPD) test OR Two well-characterized, disease-causing genetic mutations in the CF transmembrane conductance regulator (CFTR) gene AND 1 or more accompanying clinical features consistent with CF
* FEV1 ≥ 40% and ≤ 90% predicted
* BMI ≥ 19 and ≤ 30 kg/m2
* Clinically stable with no evidence of significant new or acute respiratory symptoms
* Chest radiograph without significant acute findings; or chest radiograph, CT, or MRI obtained and interpreted within 90 days prior to enrollment, without acute findings and no significant intercurrent illness; chronic, stable findings are allowed
* History of lifetime smoking < 5 pack-years (ie, 1 pack per day x 1 year =

  1 pack-year) and non-smokers of at least 60 days duration prior to Screening
* Estimated creatinine clearance ≥ 80 mL/min at Screening
* Negative drug tests; including alcohol
* Hepatitis B, C, & HIV Negative
* Surgically sterile or ≥ 12 months post-menopausal
* Non-pregnant females

Exclusion Criteria:

* Experienced symptoms of recent acute upper or lower respiratory tract infection or acute pulmonary exacerbation requiring treatment within 2 weeks prior to Screening
* Plasma potassium ≥ 5 mEq/L
* Changes in chronic azithromycin use, bronchodilator (BD), dornase alfa, HS, physiotherapy technique or regimen, antibiotics or corticosteroid medications within 28 days prior to Screening
* History of sputum or throat swab culture yielding Burkholderia species within 2 years of Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of GS-5737 | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Compass Research Phase 1, LLC, Orlando, Florida, United States